CLINICAL TRIAL: NCT02047656
Title: A Two Part Study Including a Randomized, Double Blind, Placebo Controlled, Multiple Dose Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LFF269 After b.i.d Dosing in Healthy Volunteers and an Open Label, Multiple Dose Pharmacokinetics Study in Hypertension Subjects
Brief Title: To Evaluate Pharmacokinetics of LFF269 in Healthy Volunteers and Patients With Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLFF269X2105
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Part 1 - Healthy Volunteers; Part 2 - Patients With Hypertension
Keywords: Healthy volunteers, hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo to LFF269 (Part 1) (Placebo Comparator): Placebo to LFF269 twice daily (b.i.d) for 10 days in healthy volunteers
  Interventions: Drug: Placebo to LFF269
- LFF269 (Part 1) (Experimental): LFF269 twice daily (b.i.d) for 10 days in healthy volunteers
  Interventions: Drug: LFF269
- LFF269 (Part 2) (Experimental): LFF269 twice daily (b.i.d) for 5 days in patients with hypertension
  Interventions: Drug: LFF269

INTERVENTIONS:
Drug: LFF269 — LFF269 capsules twice daily (b.i.d)
  Other Names: LFF269 active
  Arms: LFF269 (Part 1); LFF269 (Part 2)
Drug: Placebo to LFF269 — Placebo LFF269 b.i.d for 10 days in healthy volunteers
  Other Names: placebo
  Arms: Placebo to LFF269 (Part 1)

SUMMARY:
This study is designed to enable optimal dose selection of LFF269 for potential future studies by providing additional information about the compounds safety, tolerability, pharmacokinetic and pharmacodynamic profiles.

ELIGIBILITY:
Inclusion Criteria:

Part 1

- Healthy men and women of non-childbearing potential, 18 to 80 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.

Part 2

* Hypertensive men and women of non-childbearing potential, 18 to 80 years of age inclusive.
* Patients with mild-to-moderate uncomplicated essential hypertension

Exclusion Criteria:

Part 1

* History of hypersensitivity or allergy to any of the study drugs or to drugs of similar chemical classes.
* A history of clinically significant ECG abnormalities.
* Known history or current clinically significant arrhythmias.
* History of hypertension, adrenal or endocrine disease.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant.
* Smokers (use of tobacco products in the previous 3 months).
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen or Hepatitis C test result.

Part 2

* Pregnant or nursing (lactating) women.
* Women of child-bearing potential.
* Known history or evidence of a secondary form of hypertension
* Type 1 or type 2 diabetes mellitus.
* History of heart diseases
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result.

Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Number of healthy volunteers reported with adverse events as an assessment of safety and tolerability (Part 1) | 10 days

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau)[Part 1- Healthy volunteers] | Day 1
Observed maximum plasma concentration following drug administration (Cmax) at day 1 [Part 1- Healthy volunteers] | Day 1
Area Under the Plasma Concentration-time Curve From Time Zero to the End of the Dosing Interval Tau (AUCtau) [Part 2- Patients with hypertension] | Day 1
Observed maximum plasma concentration following drug administration (Cmax) at day 1 [Part 2 - Patients with hypertension] | Day 1
Area under the plasma concentration-time curve from time zero to the end of the dosing interval tau at steady state (AUCtau,ss) [Part 1- Healthy volunteers] | Day 10
Area under the plasma concentration-time curve from time zero to the end of the dosing interval tau at steady state (AUCtau,ss) [Part 2 - Patients with hypertension] | Day 5
Observed maximum plasma concentration following drug administration at steady state (Cmax,ss) [Part 2 - Patients with hypertension] | Up to Day 5
Observed maximum plasma concentration following drug administration at steady state (Cmax,ss) [Part 1- Healthy volunteers] | Up to Day 10
Number of patients reported with adverse events as an assessment of safety and tolerability (Part - 2, Patient with Hypertension) | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Miami, Florida, United States